CLINICAL TRIAL: NCT01509638
Title: A Pain Relief Trial Utilizing the Infiltration of a Multivesicular Liposome Formulation Of Bupivacaine, EXPAREL®: A Phase 4 Health Economic Trial in Adult Patients Undergoing Ileostomy Reversal
Brief Title: A Health Economic Trial in Adult Patients Undergoing Ileostomy Reversal MA402S23B501
Acronym: IMPROVE-IR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Collaborators: Registrat-Mapi (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MA402S23B501
Record Dates: First submitted 2011-10-24; First posted 2012-01-13 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-01

CONDITIONS: Retraction of Colostomy
Keywords: Ileostomy reversal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Standard of Care (Active Comparator): IV Morphine sulfate or Sponsor-approved equivalent via a patient-controlled analgesia (PCA) pump
  Interventions: Drug: Group 1 Standard of Care
- Group 2 EXPAREL (Active Comparator): bupivacaine liposome injectable suspension.
  Interventions: Drug: Group 2 EXPAREL

INTERVENTIONS:
Drug: Group 1 Standard of Care — Patients in this group will receive IV morphine sulfate or Sponsor-approved equivalent via PCA pump, as needed.
  Arms: Group 1 Standard of Care
Drug: Group 2 EXPAREL — Patients in this group will receive 266 mg EXPAREL diluted with preservative-free 0.9% normal saline to a total volume of 30cc and administered via wound infiltration prior to wound closure. When not contraindicated, 30 mg IV ketorolac will be given at the end of surgery. If not indicated, IV non-steroidal anti-inflammatory drug (NSAID) may be substituted per the site's standard of care.
  Other Names: bupivacaine liposome injectable suspension
  Arms: Group 2 EXPAREL

SUMMARY:
This study is designed to compare the standard of care against EXPAREL (bupivacaine liposome injectable suspension) to determine if total opioid consumption is reduced when using EXPAREL, therefore possibly reducing total hospitalization costs.

DETAILED DESCRIPTION:
This is a phase 4, prospective, sequential, open-label study designed to evaluate the efficacy, safety, and health economic benefits of intraoperative local wound infiltration with EXPAREL (bupivacaine liposome injectable suspension) compared with postsurgical administration of standardized intravenous (IV) morphine sulfate or Sponsor-approved equivalent for postsurgical analgesia in adult patients undergoing ileostomy reversal with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Patients scheduled to undergo ileostomy reversal.
* Ability to provide informed consent, adhere to study visit schedule, and complete all assessments.

Exclusion Criteria:

* Patients with a history of hypersensitivity or idiosyncratic reactions or intolerance to any local anesthetic, opioid, or propofol.
* Patients who abuse alcohol or other drug substance.
* Patients with severe hepatic impairment.
* Patients currently pregnant or who may become pregnant during the course of the study or who are unwilling to use acceptable means of contraception for at least one month before and one month after dosing.
* Patients with any psychiatric, psychological, or other condition that the Investigator feels may make the patient an inappropriate candidate for this clinical study.
* Patients who have participated in an EXPAREL study within the last 30 days.
* Patients who have received an investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during the patient's participation in this study.

In addition, the patient will be ineligible if he/she meets the following criteria during surgery:

* Patients who have any concurrent surgical procedure.
* Patients who receive intraoperative administration of opioids (other than fentanyl or analogs) or any other analgesic, local anesthetics, or anti-inflammatory agents.
* Patients who receive Entereg(R).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marylise Boutros, M.D., Principal Investigator — Cleveland Clinic Florida
Locations (2):
- United States (2):
  - Cleveland Clinic Florida, Weston, Florida
  - Cleveland Clinic Ohio, Beachwood, Ohio

REFERENCES:
- [Derived] Cohen SM, Vogel JD, Marcet JE, Candiotti KA. Liposome bupivacaine for improvement in economic outcomes and opioid burden in GI surgery: IMPROVE Study pooled analysis. J Pain Res. 2014 Jun 24;7:359-66. doi: 10.2147/JPR.S63764. eCollection 2014. PMID 25018650

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 patients in Group 1 and 25 patients in Group 2 were enrolled. 22 patients from Group 1 and 23 patients from Group 2 were in the Safety Analysis Set (patients who underwent planned surgery). Efficacy Analysis Set was 20 patients from Group 1 and 23 from Group 2 (planned surgery, no exclusion criteria, informed consent, Group 2 received EXPAREL)
Period: Overall Study
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL
Started | 23 | 26
Completed | 20 | 24
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Population: 23 patients in Group 1 and 25 patients in Group 2 were enrolled. 22 patients from Group 1 and 23 patients from Group 2 were in the Safety Analysis Set (patients who underwent planned surgery).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL | Total
Number analyzed (Participants) | 22 | 25 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (17.87) | 48.2 (14.53) | 47.7 (16.01)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 24 | 42
  >=65 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  United States | 22 | 25 | 47

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Burden
Description: Total opioid consumed (IV and PO) postsurgically until hospital discharge order is written or through Day 30, whichever is sooner.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner
Population: 22 patients from Group 1 and 25 patients from Group 2 were in the Safety Analysis Set (patients who underwent planned surgery). Efficacy Analysis Set was 20 patients from Group 1 and 23 from Group 2 (planned surgery, no exclusion criteria, informed consent, Group 2 received EXPAREL)
Measure: Mean (Standard Deviation); unit: mg morphine equivalent
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL
Number analyzed (Participants) | 20 | 23
mg morphine equivalent | 67.7 (46.64) | 38.41 (45.85)

2. Primary Outcome: Health Economic Benefits
Description: Total cost of hospitalization until the time the discharge order is written or through Day 30, whichever is sooner.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL
Number analyzed (Participants) | 20 | 23
dollars | 7284.63 (3577.42) | 7010.16 (2709.56)

3. Primary Outcome: Health Economic Benefit
Description: Length of stay (LOS), recorded in hours, defined as the time of completion of the wound closure until the hospital discharge order is written or through Day 30, whichever is sooner.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL
Number analyzed (Participants) | 20 | 23
days | 4 [2 to 7] | 3 [1 to 15]

4. Secondary Outcome: Incidence of Opioid-related Adverse Events
Description: Incidence of opioid-related adverse events defined as somnolence, respiratory depression, hypoventilation, hypoxia, dry mouth, nausea, vomiting, constipation, sedation, confusion, pruritus, urinary retention, and postoperative ileus.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL
Number analyzed (Participants) | 20 | 23
number of events | 0.1 (0.22) | 0.1 (0.29)

5. Secondary Outcome: Patient Satisfaction With Postsurgical Analgesia
Description: Responses to one question pertaining to patient satisfaction with postsurgical analgesia
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: Efficacy Analysis Set was 20 patients from Group 1 and 23 from Group 2 (planned surgery, no exclusion criteria, informed consent, Group 2 received EXPAREL)
Measure: Number; unit: participants
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL
Number analyzed (Participants) | 20 | 23
participants
  Extremely Satisfied | 8 | 11
  Satisified | 7 | 9
  Neither Satisfied nor Dissatisfied | 1 | 2
  Dissatisfied | 0 | 1
  Not Reported | 4 | 0

6. Secondary Outcome: Patient Discharged From Hospital for at Least 3 Days
Description: Yes, if patient discharged from hospital for at least 3 days; no, if patient not discharged from hospital for at least 3 day; not reported, if applicable.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL
Number analyzed (Participants) | 20 | 23
participants | 16 | 22

7. Secondary Outcome: Patient Made Unplanned Visit(s) With Any Healthcare Providers
Description: Yes, if patient made unplanned visit(s); No, if patient did not make unplanned visits; not reported, if applicable
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 5
Measure: Number; unit: participants who answered yes
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL
Number analyzed (Participants) | 20 | 23
participants who answered yes | 2 | 4

8. Secondary Outcome: Contact or Attempted to Contact Surgeon/Doctor to Discuss Recovery After Surgery
Description: Yes, if contacted or attempted to contact; No, if did not contact and did not attempt to contact; not reported, if applicable.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 5
Measure: Number; unit: participants who answered yes
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL
Number analyzed (Participants) | 20 | 23
participants who answered yes | 5 | 2

9. Secondary Outcome: Experienced Health Problems or Changes in Health Since Hospital Discharge
Description: Yes, if experienced health problems or changes in health; No, if did not experience health problems or changes in health; not reported, if applicable
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 5
Measure: Number; unit: participants who answered yes
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL
Number analyzed (Participants) | 20 | 23
participants who answered yes | 4 | 5

10. Secondary Outcome: Time to First Opioid Administration
Description: Time in hours to first opioid administration
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL
Number analyzed (Participants) | 20 | 23
hours | 0.7 [0.3 to 3.6] | 1.1 [0.3 to 71]

ADVERSE EVENTS:
Time Frame: 30 days post surgery
Description: Normal systematic assessment of adverse events. 22 patients from Group 1 and 25 patients from Group 2 were in the Safety Analysis Set (patients who underwent planned surgery).
Arm/Group | Group 1 Standard of Care | Group 2 EXPAREL
Serious Adverse Events (participants affected / at risk) | 0/22 | 3/25
Other Adverse Events (participants affected / at risk) | 18/22 | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Standard of Care (N=22) | Group 2 EXPAREL (N=25)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (Immune system disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Anastomatic complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Standard of Care (N=22) | Group 2 EXPAREL (N=25)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyoderma gangrinosum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema peripheral (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 1 (1)
Postprocedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No